CLINICAL TRIAL: NCT06875284
Title: Evaluating Cross-Cutting Sexual Assault and Alcohol Misuse Prevention Programming at the U.S. Air Force Academy
Brief Title: Evaluating Cross-Cutting Prevention at the U.S. Air Force Academy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency); University of Florida (Other); San Diego State University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marni Kan, Senior Prevention Researcher, RTI International
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0218275.001.001.003; W81XWH-21-9-0011.012 (Other Grant/Funding Number: U.S. Army Medical Research and Development Command); W81XWH-20-2-0014 (Other Grant/Funding Number: The Department of Defense's Office of Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2025-03-03; First posted 2025-03-13 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Sexual Assault; Alcohol Misuse
Keywords: Sexual assault prevention; Alcohol misuse prevention; Sexual Communication and Consent; eCHECKUP TO GO
MeSH Terms: interventions — Consent Forms; Ethanol

STUDY DESIGN:
Intervention Model Description: Quasi-experimental trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Training as usual (TAU) (Active Comparator): TAU without SCC or eCHECKUP TO GO
  Interventions: Behavioral: Training as usual (TAU)
- TAU plus eCHECKUP TO GO (Experimental): TAU with eCHECKUP TO GO (without SCC)
  Interventions: Behavioral: Alcohol eCHECKUP TO GO (eCHECKUP TO GO); Behavioral: Training as usual (TAU)
- SCC (Experimental): SCC without TAU or eCHECKUP TO GO
  Interventions: Behavioral: Sexual Communication and Consent (SCC)
- SCC plus eCHECKUP TO GO (Experimental): SCC with eCHECKUP TO GO (without TAU)
  Interventions: Behavioral: Sexual Communication and Consent (SCC); Behavioral: Alcohol eCHECKUP TO GO (eCHECKUP TO GO)

INTERVENTIONS:
Behavioral: Sexual Communication and Consent (SCC) — SCC combines universal classroom instruction with tailored web-based content. Based on sociodemographic characteristics and prior sexual assault experiences, Cadets receive tailored content that addresses either primary victimization prevention, revictimization prevention, or healthy relationships and bystander intervention promotion.
  Arms: SCC; SCC plus eCHECKUP TO GO
Behavioral: Alcohol eCHECKUP TO GO (eCHECKUP TO GO) — eCHECKUP TO GO is a personalized, online intervention designed to reduce cognitive risk factors for alcohol misuse. eCHECKUP TO GO is brief, self-guided, and provides individualized feedback based on a user's self-reported alcohol use patterns and consequences.
  Arms: SCC plus eCHECKUP TO GO; TAU plus eCHECKUP TO GO
Behavioral: Training as usual (TAU) — TAU involves universal classroom instruction focused on developing knowledge, attitudes, and skills to promote personal resilience, increase potential for success, and develop healthy and rewarding personal relationships.
  Arms: TAU plus eCHECKUP TO GO; Training as usual (TAU)

SUMMARY:
Sexual assault and alcohol misuse are interrelated, persist at high rates in military populations, and carry negative consequences for military units and personnel. Combining tailored efforts to prevent sexual assault and alcohol misuse is critical for developing a more effective Force. This study will test the cross-cutting immediate and long-term outcomes of two programs, the Sexual Communication and Consent (SCC) sexual assault prevention program and the eCHECKUP TO GO alcohol misuse prevention program, delivered separately and in combination, with Cadets at the United States Air Force Academy. Anonymous Cadet self-report data will be collected before training (pre-test), immediately after training (post-test), 3 months after training (Fall semester follow-up), and 9 months after training (Spring semester follow-up).

DETAILED DESCRIPTION:
Sexual assault and alcohol misuse both persist at high rates among military populations. These behaviors interfere with readiness, unit cohesion, mission objectives, and personnel performance and retention. There are demonstrated associations between sexual assault and alcohol misuse for both perpetrators and victims of sexual assault. Therefore, combining efforts to prevent sexual assault and alcohol misuse is critical for more effective and efficient programming. Moreover, tailored prevention programming that addresses individual risks and experiences related to sexual assault and alcohol misuse is likely to be the most effective programming. Unfortunately, to date, no evidence-based cross-cutting interventions have been developed and evaluated for impacts on both sexual assault and alcohol misuse among military populations. Several challenges impede this effort. Sexual assault prevention and alcohol misuse prevention are typically managed in different organizations within military settings, including within Military Service Academies. Training settings face many competing demands for trainees' time and instructor capacity, and instructors' ability to provide both sexual assault-related and alcohol-related training varies widely. Despite the promise of tailored training, individualized programming also presents feasibility challenges in group education settings common to military training. In alignment with the Fiscal Years 2021-2025 Department of Defense (DoD) Sexual Assault Prevention and Response (SAPR) Research Agenda and DoD's desire to have cross-cutting prevention programs that reduce risk for multiple harmful behaviors, the long-term goal of the proposed work is to address these challenges and provide the military with flexible, engaging, tailored prevention programming that reduces sexual assault and alcohol misuse while minimizing burden on Service members and training settings. To that end, the basic objective of this study is to test the cross-cutting immediate and long-term outcomes of two programs, the Sexual Communication and Consent (SCC) sexual assault prevention program and the eCHECKUP TO GO alcohol misuse prevention program, delivered separately and in combination, with Cadets at the United States Air Force Academy. Anonymous Cadet self-report data will be collected before training (pre-test), immediately after training (post-test), 3 months after training (Fall semester follow-up), and 9 months after training (Spring semester follow-up).

ELIGIBILITY:
Inclusion Criteria:

* U.S. Air Force Academy Basic Cadet enrolled in 2022 or 2023 Basic Cadet Training

Exclusion Criteria:

* Unable or unwilling to provide informed consent

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2041 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marni L Kan, PhD, Principal Investigator — RTI International; Nichole M Scaglione, PhD, Principal Investigator — University of Florida; Emily A Schmied, PhD, Principal Investigator — San Diego State University
Locations (1):
- United States Air Force Academy, Air Force Academy, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldstein SJ, Scaglione NM, Kan ML, Grimes KEL, Lane ME, Morgan JK, Martin SL. Accuracy, Acceptability, and Burden of an Integrated Screening Approach to Facilitate the Delivery of Tailored Sexual Assault Prevention in the U.S. Air Force. J Child Sex Abus. 2025 Jul-Aug;34(5-6):661-681. doi: 10.1080/10538712.2024.2364792. Epub 2024 Jun 14. PMID 38874411
- [Background] Eckhoff R, Boyce M, Watkins RL, Kan M, Scaglione N, Pound L, Root M. Examining the Use of Mobile Technology to Deliver Tailored Sexual Assault Prevention in a Classroom Environment in the Military: Development and Usability Study. JMIR Mhealth Uhealth. 2022 Nov 16;10(11):e41455. doi: 10.2196/41455. PMID 36383404
- [Background] Kan ML, Scaglione NM, Buben A, Morgan JK, Grimes KEL, Watson CJ, Charm S, Lowe AN, Eckhoff RP, Lane M, Root MK, Pound LB. Feasibility and acceptability of tailored sexual assault prevention in the US Air Force. Pilot Feasibility Stud. 2024 Nov 21;10(1):145. doi: 10.1186/s40814-024-01565-6. PMID 39574150

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Squadrons
Groups:
- Sexual Communication and Consent (SCC): SCC without TAU or eCHECKUP TO GO
  Sexual Communication and Consent (SCC): SCC combines universal classroom instruction with tailored web-based content. Based on sociodemographic characteristics and prior sexual assault experiences, Cadets receive tailored content that addresses either primary victimization prevention, revictimization prevention, or healthy relationships and bystander intervention promotion.
Period: Overall Study
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Started (To be counted as having started this study, participants must have provided any outcome measure data during the pretest assessment window (validated based on survey completion timestamp) and consented to the use of survey data for research purposes.) | 556; 5 Squadrons | 401; 3 Squadrons | 632; 5 Squadrons | 396; 3 Squadrons
Posttest (To be counted as having participated in the posttest assessment for this study, participants must have provided any outcome measure data during the posttest assessment window (validated based on survey completion timestamp) and consented to the use of survey data for research purposes.) | 560; 5 Squadrons | 328; 3 Squadrons | 490; 5 Squadrons | 337; 3 Squadrons
3-month follow-up (To be counted as having participated in this assessment, participants must have provided any outcome measure data during the 3-month follow-up assessment window (validated based on survey completion timestamp) and consented to the use of survey data for research purposes.) | 89; 5 Squadrons | 21; 3 Squadrons | 94; 5 Squadrons | 28; 3 Squadrons
Completed (To be counted as having completed this study, participants must have provided any outcome measure data during the 9-month follow-up assessment window (validated based on survey completion timestamp) and consented to the use of survey data for research purposes.) | 24; 5 Squadrons | 13; 3 Squadrons | 31; 5 Squadrons | 11; 3 Squadrons
Not Completed | 532; 0 Squadrons | 388; 0 Squadrons | 601; 0 Squadrons | 385; 0 Squadrons

BASELINE CHARACTERISTICS:
Groups:
- Sexual Communication and Consent (SCC): Sexual Communication and Consent without TAU or eCHECKUP TO GO
- Total: Total of all reporting groups
Arm/Group | Training as Usual (TAU) | TAU Plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC Plus eCHECKUP TO GO | Total
Number analyzed (Participants) | 556 | 401 | 632 | 396 | 1985
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.33 (0.98) | 18.35 (0.86) | 18.29 (0.93) | 18.34 (0.91) | 18.32 (0.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 118 | 173 | 107 | 554
  Male | 400 | 283 | 459 | 289 | 1431
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 45 | 38 | 54 | 37 | 174
  Black or African American | 30 | 14 | 32 | 16 | 92
  Native American or Alaska Native | 1 | 0 | 1 | 0 | 2
  Pacific Islander/Native Hawaiian | 1 | 1 | 6 | 0 | 8
  Spanish/Hispanic/Latino/a | 64 | 39 | 64 | 38 | 205
  White | 345 | 262 | 396 | 263 | 1266
  Multiple races/ethnicities | 63 | 38 | 61 | 32 | 194
  Prefer not to answer or missing | 5 | 9 | 14 | 6 | 34
  Other race/ethnicity | 2 | 0 | 4 | 4 | 10
Self-reported Sexual Assault Victimization [Count of Participants; unit: Participants] — Participants self-report whether they experienced any type of unwanted sexual contact prior to arriving at USAFA to begin Basic Cadet Training.
  Participants | 88 | 63 | 92 | 69 | 312
Self-reported Sexual Assault Perpetration [Count of Participants; unit: Participants] — Participants self-report whether they perpetrated any type of unwanted sexual contact prior to arriving at USAFA to begin Basic Cadet Training.
  Participants | 6 | 6 | 8 | 7 | 27
Self-reported Alcohol Use [Count of Participants; unit: Participants] — Participants self-report the approximate number of alcoholic drinks they consumed each day of the week during a typical week over the past month. Participants who respond with any weekly value greater than 0 alcoholic drinks at either the Fall or Spring semester follow-up are coded as positive for any alcohol use.
  Participants | 122 | 93 | 130 | 89 | 434

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Sexual Assault Victimization
Description: Participants self-report whether they experienced any type of unwanted sexual contact between Basic Cadet Training and the Spring semester follow-up using a modified version of the Sexual Experiences Survey.
Time Frame: From pre-test to Spring semester follow-up, an average of 10 months
Population: The number analyzed at follow-up differs from the overall number analyzed because not all participants who provided pre-test data provided follow-up data.
Measure: Count of Participants; unit: Participants
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Number analyzed (Participants) | 556 | 401 | 632 | 396
Participants
  Pretest | 88 | 63 | 92 | 69
  9-month follow-up: number analyzed (Participants) | 24 | 13 | 31 | 11
  9-month follow-up | 1 | 0 | 0 | 0

2. Primary Outcome: Self-reported Sexual Assault Perpetration
Description: Participants self-report whether they perpetrated any type of unwanted sexual contact between Basic Cadet Training and the Spring semester follow-up using a modified version of the Sexual Experiences Survey.
Time Frame: From pre-test to Spring semester follow-up, an average of 10 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Number analyzed (Participants) | 556 | 401 | 632 | 396
Participants
  Pretest | 6 | 6 | 8 | 7
  9-month follow-up: number analyzed (Participants) | 24 | 13 | 31 | 11
  9-month follow-up | 0 | 0 | 0 | 0

3. Primary Outcome: Self-reported Alcohol Use
Description: Participants self-report the approximate number of alcoholic drinks they consumed each day of the week during a typical week over the past month (assessed at both the Fall and Spring semester follow-up assessments). Participants who respond with any weekly value greater than 0 alcoholic drinks at either the Fall or Spring semester follow-up are coded as positive for any alcohol use.
Time Frame: From pre-test to Spring semester follow-up, an average of 10 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Number analyzed (Participants) | 556 | 401 | 632 | 396
Participants
  Pretest | 122 | 93 | 130 | 89
  9-month follow-up: number analyzed (Participants) | 24 | 13 | 31 | 11
  9-month follow-up | 18 | 5 | 14 | 9

4. Secondary Outcome: Knowledge of Sexual Assault
Description: The percentage of correct participant responses to 8 true-or-false questions about sexual assault.
Time Frame: From pre-test to post-test, an average of 1 month
Population: The number analyzed at post-test differs from the overall number analyzed because not all participants who provided pre-test data provided post-test data.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Number analyzed (Participants) | 549 | 399 | 621 | 396
percentage of correct responses
  Pretest value | 78.10 (14.61) | 76.53 (15.33) | 78.97 (14.55) | 78.30 (15.16)
  Posttest value: number analyzed (Participants) | 545 | 326 | 481 | 333
  Posttest value | 82.74 (13.66) | 81.85 (13.57) | 90.79 (11.01) | 92.32 (10.11)
Statistical Analysis 1: Comparison: Training as usual (TAU) vs SCC plus eCHECKUP TO GO; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -9.01, 95% CI 2-sided [-11.06 to -6.96], Standard Error of Mean 1.05 — The SCC plus eCHECKUP TO GO arm was the reference group
Statistical Analysis 2: Comparison: Sexual Communication and Consent (SCC) vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.041, Mixed Models Analysis; Mean Difference (Net) = -2.16, 95% CI 2-sided [-4.22 to -0.09], Standard Error of Mean 1.05 — The SCC plus eCHECKUP TO GO arm was the reference group
Statistical Analysis 3: Comparison: TAU plus eCHECKUP TO GO vs SCC plus eCHECKUP TO GO; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -8.51, 95% CI 2-sided [-10.76 to -6.25], Standard Error of Mean 1.15 — Covariates included cohort and history of peer victimization; The SCC plus eCHECKUP TO GO arm was the reference group

5. Secondary Outcome: Knowledge of Effective Consent
Description: The percentage of correct participant responses to 7 true-or-false questions about effective sexual consent.
Time Frame: From pre-test to post-test, an average of 1 month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Number analyzed (Participants) | 546 | 396 | 622 | 395
percentage of correct responses
  Pretest value | 96.64 (6.99) | 96.86 (6.58) | 96.37 (7.42) | 96.45 (6.96)
  Posttest value: number analyzed (Participants) | 538 | 321 | 465 | 332
  Posttest value | 97.57 (5.89) | 97.57 (5.95) | 98.16 (4.93) | 98.53 (4.57)
Statistical Analysis 1: Comparison: Training as usual (TAU) vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.035, Mixed Models Analysis; Mean Difference (Net) = -1.18, 95% CI 2-sided [-2.27 to -0.08], Standard Error of Mean 0.56 — The SCC plus eCHECKUP TO GO arm was the reference group
Statistical Analysis 2: Comparison: Sexual Communication and Consent (SCC) vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.54, Mixed Models Analysis; Mean Difference (Net) = -0.34, 95% CI 2-sided [-1.44 to 0.76], Standard Error of Mean 0.56 — The SCC plus eCHECKUP TO GO arm was the reference group
Statistical Analysis 3: Comparison: TAU plus eCHECKUP TO GO vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.023, Mixed Models Analysis; Mean Difference (Net) = -1.40, 95% CI 2-sided [-2.60 to -0.19], Standard Error of Mean 0.61

6. Secondary Outcome: Self-efficacy to Resist Unwanted Sexual Advances
Description: A subset of participants rate their degree of confidence in their ability to use certain protective strategies in 6 specific high-risk situations. Scale scores range 6 to 42, with higher scores indicating greater self-efficacy.
Time Frame: From pre-test to post-test, an average of 1 month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Number analyzed (Participants) | 178 | 137 | 194 | 121
score on a scale
  Pretest value | 33.45 (5.91) | 33.45 (7.00) | 33.11 (5.68) | 32.05 (7.05)
  Posttest value: number analyzed (Participants) | 172 | 108 | 141 | 103
  Posttest value | 34.68 (6.04) | 34.75 (6.58) | 34.84 (5.45) | 35.96 (5.50)
Statistical Analysis 1: Comparison: Training as usual (TAU) vs SCC plus eCHECKUP TO GO; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -2.66, 95% CI 2-sided [-3.98 to -1.34], Standard Error of Mean 0.67 — The SCC plus eCHECKUP TO GO arm was the reference group
Statistical Analysis 2: Comparison: Sexual Communication and Consent (SCC) vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.012, Mixed Models Analysis; Mean Difference (Net) = -1.74, 95% CI 2-sided [-3.09 to -0.39], Standard Error of Mean 0.69 — The SCC plus eCHECKUP TO GO arm was the reference group
Statistical Analysis 3: Comparison: TAU plus eCHECKUP TO GO vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Median Difference (Net) = -2.45, 95% CI 2-sided [-3.88 to -1.03], Standard Error of Mean 0.73 — The SCC plus eCHECKUP TO GO arm was the reference group

7. Secondary Outcome: Normative Perceptions of Peer Alcohol Use
Description: Participants report how many days in the week they estimate the average Cadet of their same age and gender drinks and how many drinks the average Cadet of their same age and gender consumes per day using a modified version of the Quantity/Frequency/Peak questionnaire. The average number of estimated drinks consumed per drinking day is computed from this data and has a possible score range of 0 drinks to 6 drinks.
Time Frame: From pre-test to post-test, an average of 1 month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Number analyzed (Participants) | 508 | 374 | 590 | 369
score on a scale
  Pretest value | 2.89 (3.69) | 2.67 (3.50) | 3.11 (3.81) | 2.66 (3.30)
  Posttest value: number analyzed (Participants) | 495 | 289 | 390 | 308
  Posttest value | 3.69 (4.17) | 2.52 (3.09) | 2.72 (3.53) | 2.88 (3.05)
Statistical Analysis 1: Comparison: Training as usual (TAU) vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.058, Mixed Models Analysis; Mean Difference (Net) = 0.50, 95% CI 2-sided [-0.02 to 1.02], Standard Error of Mean 0.26 — The SCC plus eCHECKUP TO GO arm was the reference group
Statistical Analysis 2: Comparison: Sexual Communication and Consent (SCC) vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.046, Mixed Models Analysis; Mean Difference (Net) = -0.54, 95% CI 2-sided [-1.07 to -0.01], Standard Error of Mean 0.27 — The SCC plus eCHECKUP TO GO arm was the reference group
Statistical Analysis 3: Comparison: TAU plus eCHECKUP TO GO vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.097, Mixed Models Analysis; Mean Difference (Net) = -0.48, 95% CI 2-sided [-1.06 to 0.09], Standard Error of Mean 0.29 — The SCC plus eCHECKUP TO GO arm was the reference group

8. Secondary Outcome: Readiness to Change Alcohol Use Behavior
Description: Participants self-report their readiness to change their drinking behavior using a single item. The possible item score ranges 0 to 4, with higher scores indicating greater readiness to change.
Time Frame: From pre-test to post-test, an average of 1 month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Number analyzed (Participants) | 421 | 345 | 492 | 343
score on a scale
  Pretest value | 0.87 (1.36) | 1.04 (1.40) | 1.02 (1.44) | 0.94 (1.39)
  Posttest value: number analyzed (Participants) | 399 | 276 | 372 | 302
  Posttest value | 1.11 (1.48) | 0.88 (1.37) | 1.28 (1.51) | 1.09 (1.43)
Statistical Analysis 1: Comparison: Training as usual (TAU) vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.64, Mixed Models Analysis; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.16 to 0.26], Standard Error of Mean 0.11 — The SCC plus eCHECKUP TO GO arm was the reference group
Statistical Analysis 2: Comparison: Sexual Communication and Consent (SCC) vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.25, Mixed Models Analysis; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.09 to 0.33], Standard Error of Mean 0.11 — The SCC plus eCHECKUP TO GO arm was the reference group
Statistical Analysis 3: Comparison: TAU plus eCHECKUP TO GO vs SCC plus eCHECKUP TO GO; Test type: Superiority; p = 0.033, Mixed Models Analysis; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.47 to -0.02], Standard Error of Mean 0.11 — The SCC plus eCHECKUP TO GO arm was the reference group

9. Secondary Outcome: Dating-related Protective Strategy Use
Description: Participants self-report the degree to which they engaged in behavioral strategies to reduce sexual assault risk using the Dating Self-Protection Against Rape Scale. Scores range 0 to 70, with higher scores indicating greater engagement in dating-related protective behavioral strategies.
Time Frame: From pre-test to Spring semester follow-up, an average of 10 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Number analyzed (Participants) | 170 | 133 | 187 | 114
score on a scale
  Pretest | 42.23 (13.40) | 42.05 (14.82) | 40.28 (16.28) | 42.43 (14.21)
  9-month follow-up: number analyzed (Participants) | 20 | 11 | 18 | 7
  9-month follow-up | 39.5 (16.41) | 40.55 (20.04) | 37.57 (22.22) | 42.00 (17.59)

10. Secondary Outcome: Alcohol-related Protective Strategy Use
Description: Participants self-report the degree to which they engaged in behavioral strategies to reduce alcohol-related harms using an adapted version of the Protective Behavioral Strategies Survey. Scores range 0 to 100, with higher scores indicating greater engagement in alcohol-related protective strategies.
Time Frame: From pre-test to Spring semester follow-up, an average of 10 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
Number analyzed (Participants) | 430 | 367 | 501 | 356
score on a scale
  Pretest | 60.64 (30.65) | 63.34 (31.52) | 58.93 (33.22) | 64.67 (31.21)
  9-month follow-up: number analyzed (Participants) | 19 | 12 | 15 | 8
  9-month follow-up | 68.92 (28.65) | 66.77 (38.96) | 55.61 (43.06) | 73.52 (32.50)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Training as usual (TAU) | TAU plus eCHECKUP TO GO | Sexual Communication and Consent (SCC) | SCC plus eCHECKUP TO GO
All-Cause Mortality (participants affected / at risk) | 0/556 | 0/401 | 0/632 | 0/396
Serious Adverse Events (participants affected / at risk) | 0/556 | 0/401 | 0/632 | 0/396
Other Adverse Events (participants affected / at risk) | 0/556 | 0/401 | 0/632 | 0/396

LIMITATIONS AND CAVEATS:
Follow-up survey participation rates were low across all arms, therefore statistical analyses involving follow-up data were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT06875284/Prot_SAP_000.pdf